CLINICAL TRIAL: NCT05022368
Title: Surgical Safety Device Use During Transoral Surgery
Brief Title: Oral Device Clinical Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Zotarix LLC (Unknown)
Responsible Party: Principal Investigator, Tendy Chiang, Assistant professor, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000722
Record Dates: First submitted 2021-08-25; First posted 2021-08-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Tonsil Disease; Dental Diseases; Adenoid; Disorder (and Tonsils)
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Oral Safety Device (Experimental): patients on which the device "LabraGuard" is used.
  Interventions: Device: LabraGuard

INTERVENTIONS:
Device: LabraGuard — Protection of the lips and the oral commissure during transoral procedures

SUMMARY:
The investigators are studying the use of a new medical device developed at Nationwide Children's. This technology has been licensed and produced by Zotarix LLC, a medical device company. It is designed to aid in retraction and provide protection of the lips during surgery. The investigators are not recording any of your identifiable personal health information except for the surgery date. This device, called the LabraGuard is a sterile, soft medical grade silicone, and no alternative device with these exact protective properties exists, and the investigators are trying to learn more about how it performs in different age children.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 21 years of age and under
* Having a surgical procedure done through the mouth where the lips are at risk of injury
* Performed by attendings from either the Otolaryngology department or the Dental department.
* Subject/Subject's guardian provides consent to be in the study

Exclusion Criteria:

* Allergy to silicone
* Unable to achieve good fit

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Field Visibility | baseline
  Surgeons level of visibility of the oropharynx on a scale of 1 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No